CLINICAL TRIAL: NCT02361827
Title: The Effect of Vitamin D on in Vitro Fertilization Outcome, a Prospective Observational Study
Brief Title: The Effect of Vitamin D on in Vitro Fertilization Outcome
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Luoyang maternal and child hospital (Unknown)
Responsible Party: Principal Investigator, Yingpu Sun, Director of Reproductive Medicine Center, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: RMCZZU-Vitamin D
Record Dates: First submitted 2015-02-08; First posted 2015-02-12 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Ongoing Pregnancy Rate; Vitamin D; In Vitro Fertilization
Keywords: Vitamin D; IVF outcome
MeSH Terms: interventions — Embryo Transfer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum/follicle fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- A1, Vitamin D deficient: Vitamin D level before cycle < 20 ng/mL.
  Interventions: Procedure: Embryo transfer
- B1, Vitamin D insufficient: Vitamin D level before cycle 20-29.9 ng/mL
  Interventions: Procedure: Embryo transfer
- C1, Vitamin D replete: Vitamin D level before cycle > 30 ng/mL
  Interventions: Procedure: Embryo transfer
- A2, Vitamin D deficient: Vitamin D level before ET < 20 ng/mL (FET with Euploid embryos)
  Interventions: Procedure: Embryo transfer
- B2, Vitamin D insufficient: Vitamin D level before ET 20-29.9 ng/mL (FET with Euploid embryos)
  Interventions: Procedure: Embryo transfer
- C2, Vitamin D replete: Vitamin D level before ET > 30 ng/mL (FET with Euploid embryos)
  Interventions: Procedure: Embryo transfer

INTERVENTIONS:
Procedure: Embryo transfer — For patients in each group after oocyte retrieval, they will have embryo transferred 3 or 5 days after oocyte retrieval. For FET cycles, they will have ET with an euploid blastocyst.

SUMMARY:
To date, several studies have been done to explore the relationship between Vitamin D level and IVF outcome; however, the results are controversial. Sample sizes in these studies mentioned above were relatively small. In addition, there are no prospective cohort studies in this field. Thus, here the investigators carry this prospective observational cohort study to demonstrate the relationship between vitamin D level and IVF outcome.

DETAILED DESCRIPTION:
Vitamin D level is measured before the commence of IVF cycle. According to Vitamin D level, patients are divided into 3 groups: A, Deficient, <20 ng/mL; B, Insufficient, 20-29.9 ng/mL; C, Replete, >30 ng/mL.

Ongoing pregnancy rate are compared among these three groups after controlling age, number of embryos transferred, ect.

In addition, Vitamin D level is also meassured before embryo transfer in FET cycles with PGT treatment. The effect of Vitamin D on IVF outcome is detected in patients transferred with Euploid embryos.

ELIGIBILITY:
Inclusion Criteria:

1. age between 21-40 years old
2. basal FSH hormone level less than 10 mIU/mL
3. the first cycle of IVF treatment with standard long protocol
4. both ovarian present and normal uterus.

Exclusion Criteria:

1. Important data missing
2. Gametes donation cycles
3. Anyone that does not meet the inclusion criteria

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients whose IVF cycles were cancelled due to ovarian hyperstimulation syndrome were also excluded);.
Sampling Method: Probability Sample
Enrollment: 688 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks after embryo transfer
  12 weeks after embryo transfer, gestational sac with fetal heart present inside uterus

SECONDARY OUTCOMES:
Ectopic pregnancy rate | 35 days after embryo transfer
  Ectopic pregnancy is defined as serum HCG positive, yet with no gestational sac present inside uterine cavity

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqin Bu, MD, PhD, Principal Investigator — Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University
Locations (1):
- Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

REFERENCES:
- [Background] Wang K, Dong F, Ma S, Bu Z. The association between Vitamin D deficiency and clinical pregnancy rate in IVF patients with different age. Front Endocrinol (Lausanne). 2025 Jan 3;15:1485238. doi: 10.3389/fendo.2024.1485238. eCollection 2024. PMID 39829955
- [Background] Franasiak JM, Molinaro TA, Dubell EK, Scott KL, Ruiz AR, Forman EJ, Werner MD, Hong KH, Scott RT Jr. Vitamin D levels do not affect IVF outcomes following the transfer of euploid blastocysts. Am J Obstet Gynecol. 2015 Mar;212(3):315.e1-6. doi: 10.1016/j.ajog.2014.09.029. Epub 2014 Oct 11. PMID 25265402
- [Background] Fabris A, Pacheco A, Cruz M, Puente JM, Fatemi H, Garcia-Velasco JA. Impact of circulating levels of total and bioavailable serum vitamin D on pregnancy rate in egg donation recipients. Fertil Steril. 2014 Dec;102(6):1608-12. doi: 10.1016/j.fertnstert.2014.08.030. Epub 2014 Sep 23. PMID 25256926
- [Background] Paffoni A, Ferrari S, Vigano P, Pagliardini L, Papaleo E, Candiani M, Tirelli A, Fedele L, Somigliana E. Vitamin D deficiency and infertility: insights from in vitro fertilization cycles. J Clin Endocrinol Metab. 2014 Nov;99(11):E2372-6. doi: 10.1210/jc.2014-1802. Epub 2014 Aug 14. PMID 25121462
- [Background] Rudick BJ, Ingles SA, Chung K, Stanczyk FZ, Paulson RJ, Bendikson KA. Influence of vitamin D levels on in vitro fertilization outcomes in donor-recipient cycles. Fertil Steril. 2014 Feb;101(2):447-52. doi: 10.1016/j.fertnstert.2013.10.008. Epub 2013 Nov 5. PMID 24210230